CLINICAL TRIAL: NCT01574989
Title: Effects of Repetitive Transcranial Magnetic Stimulation and Transcranial DC Stimulation on Motor Function in Stroke Patients
Brief Title: Effects of rTMS and tDCS on Motor Function in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Associate Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2010-p-001461
Record Dates: First submitted 2012-02-08; First posted 2012-04-10 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Stroke; Motor Function
Keywords: direct current stimulation; magnetic stimulation; transcranial stimulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Active low-frequency rTMS/sham tDCS (Experimental): Subjects will have both the rTMS and tDCS on their scalp during the session, however only one will be active. For this arm, the rTMS will be active, low-frequency, and the tDCS will be sham. They will undergo only one session of this condition, and it will last 20 minutes.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Device: Transcranial Direct Current Stimulation (tDCS)
- Active high-frequency rTMS/sham tDCS (Experimental): Subjects will have both the rTMS and tDCS on their scalp during the session, however only one will be active. For this arm, the rTMS will be active, high-frequency, and the tDCS will be sham. They will undergo only one session of this condition, and it will last 20 minutes.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Device: Transcranial Direct Current Stimulation (tDCS)
- Sham rTMS/active anodal tDCS (Experimental): Subjects will have both the rTMS and tDCS on their scalp during the session, however only one will be active. For this arm, the tDCS will be active, anodal, and the TMS will be sham. They will undergo only one session of this condition, and it will last 20 minutes.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Device: Transcranial Direct Current Stimulation (tDCS)
- Sham rTMS/active cathodal tDCS (Experimental): Subjects will have both the rTMS and tDCS on their scalp during the session, however only one will be active. For this arm, the tDCS will be active, cathodal, and the TMS will be sham. They will undergo only one session of this condition, and it will last 20 minutes.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Device: Transcranial Direct Current Stimulation (tDCS)
- Sham rTMS/Sham tDCS (Sham Comparator): Subjects will have both the rTMS and tDCS on their scalp during the session, and both interventions will be sham. They will undergo only one session of this condition, and it will last 20 minutes.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Subjects will either undergo (1) active low-frequency rTMS (1Hz continuous), (2) active high-frequency rTMS (10Hz, 2 second trains with inter-train interval of 28 seconds) or (3) sham rTMS (using a sham coil). Each session will last 20 minutes and will be conducted at 100% of the motor threshold.
  Other Names: magnetic stimulation; Magstim
Device: Transcranial Direct Current Stimulation (tDCS) — Subjects will either undergo (1) active anodal tDCS, (2) active cathodal tDCS or (3) sham tDCS. Each session will last 20 minutes and will be conducted using 1mA with 35^2 electrodes.
  Other Names: 1x1 low-intensity direct current stimulator; Soterix Medical

SUMMARY:
In this study the investigators aim to investigate the effects of two different types of non-invasive brain stimulation techniques -- repetitive transcranial magnetic stimulation (rTMS) and transcranial direct current stimulation (tDCS) on motor function in stroke. This is a cross-over study where subjects will receive 5 sessions of stimulation (each separated by 1 week) -- with either active tDCS and sham rTMS, sham tDCS and active rTMS or both sham tDCS and rTMS.

ELIGIBILITY:
Inclusion criteria:

(1) All subjects must be between the ages of 18-90.

Exclusion criteria:

1. History of Major depression, as defined by Beck Depression scale 30;
2. Any substantial decrease in alertness, language comprehension, or attention that might interfere with understanding instructions for motor testing;
3. Contraindications to TMS

   * history of seizures
   * unexplained loss of consciousness
   * metal in the head
   * frequent or severe headaches or neck pain
   * implanted brain medical devices.
4. Contraindications to tDCS

   * metal in the head
   * implanted brain medical devices
5. Advanced liver, kidney, cardiac, or pulmonary disease;
6. A terminal medical diagnosis consistent with survival < 1 year;
7. Coexistent major neurological or psychiatric disease (to decrease number of confounders);
8. A history of significant alcohol or drug abuse in the prior 6 months;
9. Subjects may not be actively enrolled in a separate intervention study targeting stroke recovery and any other clinical trials;
10. Subjects with global aphasia and deficits of comprehension
11. Pregnancy. Female subjects of child bearing potential will be asked to take a pregnancy test. If the pregnancy test is positive, the subject may not enroll in the study.
12. Use of neuropsychotropic medications [healthy subjects only]

Additional inclusion criteria for stroke subjects:

1. First-time clinical ischemic or hemorrhagic cerebrovascular events - evidenced by a radiological (or physician's) report
2. Weakness, defined as score of less than 55 (out of 66) on arm motor Fugl-Meyer (FM) scale
3. Stroke onset >6 months prior to study enrollment .

Additional exclusion criteria for stroke subjects:

1. Subjects may not have already received TMS and/or tDCS stimulation for stroke;
2. History of epilepsy before stroke or episodes of seizures within the last six months;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Changes in cortical excitability measures | Measured for approximately 6 weeks
  We will measure cortical excitability using single- and paired-pulse transcranial magnetic stimulation (TMS) before and after each stimulation session. We will compare the measurements from before stimulation to after stimulation, in each scheduled session, as this study is measuring the effects of a single session of tDCS/rTMS.

SECONDARY OUTCOMES:
Changes in motor function | Measured for approximately 6 weeks
  We will measure motor function using behavioral tasks (ex. purdue pegboard, jebsen taylor test, range of motion) both before and after the stimulation sessions. We will compare the measurements from before stimulation to after stimulation, in each scheduled session, as this study is measuring the effects of a single session of tDCS/rTMS.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD PHD MPH, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411